CLINICAL TRIAL: NCT07017959
Title: Impact of a Human Origin Heat Inactivated Probiotics-Lactobacillus Paracasei D3.5 (LpD3.5) as Dietary Supplement on Gut Mucin and Intestinal Permeability in Adults With IBD
Brief Title: Impact of a Human Origin Heat Inactivated Probiotic-Lactobacillus Paracasei D3.5 (LpD3.5) as Dietary Supplement on Gut Mucin and Intestinal Permeability in Adults With IBD
Acronym: LIBD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Screening
Other Study IDs: STUDY008123
Record Dates: First submitted 2025-06-04; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Inflammatory Bowel Diseases
Keywords: Lactobacillus paracasei D3.5; Ulcerative colitis; Crohn's disease; Gastrointestinal symptom rating scale
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative

STUDY DESIGN:
Intervention Model Description: Participants receive one of the interventions (LpD3.5) during the initial phase of the study (for 60 days) and receive the other intervention (Placebo) during the second phase of the study
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): LpD3.5 supplementation.
  Interventions: Dietary Supplement: LpD3.5 supplementation.
- Placebo Comparator (Placebo Comparator): Placebo supplementation.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: LpD3.5 supplementation. — Dietary Supplement: LpD3.5 are in the form of capsule where LpD3.5 contains 167 mg of LpD3.5, with the remaining portion consisting of inactive ingredients like maltodextrin
  Arms: Experimental group
Dietary Supplement: Placebo — Placebo capsules contain only inactive ingredient maltodextrin
  Arms: Placebo Comparator

SUMMARY:
This study aims to study a biological phenomenon of reduced mucin barriers that are linked with increased intestinal permeabil-ity in the gut of individuals with IBD and determine whether and how a human originated, and heat inactivated probiotic LpD3.5 impact these biological mechanisms. We plan a cross-over ran-domized placebo-controlled pilot study of n=15 individuals with IBD, who will be consented with a goal for 10 participants ran-domized in placebo (n=5) and LpD3.5 (n=5) arms to complete the study and will be given two corresponding dietary supple-ment grade capsules per day of placebo or LpD3.5 (167 mg/ capsule), respectively, for 60 days. We will have a 60-day washout period, after which participants will be cross-over in opposite arms and further intervention will be monitored at 30 and 60 days. Stool and blood samples will be collected at base-line (before intervention), and after 30, and 60 days of the start of the intervention. After a 60-day washout interval, the sample collection will be performed in a crossover fashion in opposite arms. We will analyze the levels of post-intervention fecal mucin (marker of gut barriers) between LpD3.5 and placebo groups as primary outcomes. Microbiome indices and phylogenetic abun-dances, and markers of elevated gut permeability (LBP and sCD14) will be as secondary outcomes. Our exploratory out-comes will include inflammation (IL-6, TNF-α, and IL-1β in blood, and calprotectin in feces), dose and frequency of medica-tions, and QOL questionnaires.

DETAILED DESCRIPTION:
IBD is becoming more common in both developed and developing nations, putting a significant strain on the healthcare system. IBD is now a major public health problem that affects ~3.6 million people in the United States and Europe. In 2019, there were approximately 4.9 million cases of IBD worldwide, with China and the USA having the maximum number of cases (911 405 and 762 890 (66.9 and 245.3 cases per 100,000 people, respectively). Accumulating evidence suggests that an abnormal gut microbiota composition, termed as dysbiosis, plays a key role in the pathogenesis of IBDs such as ulcerative colitis (UC) and Crohn's disease (CD). Individuals with IBDs experience pain, extreme discomfort, and numerous other symptoms caused by continuously relapsing and remitting inflammatory lesions in the layer of cells that lines the intestinal lumen (mucosa). The exact causes for IBD still are poorly understood. IBD pathogenesis is perpetuated by abnormal immune responses, which are and related with abnormalities in the intestinal epithelial barrier, enteric nervous system, and changes in microbiota composition.

While anti-inflammatory medications and antibiotics can reduce acute inflammation and fight local infections during IBD flare-ups, their usage is not without consequences. Anti-inflammatory drugs can have severe side effects, and antibiotics can disrupt the beneficial parts of the microbiome. Importantly, there are no wound treatments available that could be given to inflamed lesions directly from inside the gut lumen to speed up healing and reduce the use of those drugs.

On the other hand, probiotics have shown promise in reducing the symptoms of IBD; however, probiotics therapy has limitations. For example, (1) the beneficial effects of probiotics are highly variable, and their significance in clinical settings remains elusive; and (2) probiotics are live bacteria, posing the threat of them leaking into the blood circulation, which can increase the risk of bacterial sepsis. Moreover, there is a lack of preclinical research and clinical trials on probiotics as preventive and therapeutic treatments for CD, particularly at an early age.

We recently discovered a human-origin probiotic strain called LpD3.5 which strengthens intestinal barrier functions and reduces inflammation by restoring intestinal mucus layer. We found that this strain is effective and beneficial even when heat-killed; thus, we call it a postbiotic. Postbiotics are non-viable bacterial products or metabolic byproducts produced by probiotic microorganisms that have biologic activity in the host. Their advantages over probiotics include a lower risk of infection and reducing negative effects caused by certain microorganisms. Indeed, administering live probiotics to persons with weaker immune systems may boost inflammatory reactions and change "generally recognized as safe" harmless probiotic bacteria into harmful pathogens. Hence, the postbiotics LpD3.5 strain is under production in the Good Manufacturing Practice (GMP) facilities for human consumption and will be ready for clinical use. In our previous animal studies, we showed that LpD3.5 feeding significantly increases mucin production and proportionately increases in the abundance of the mucin-degrading bacterium Akkermansia muciniphila. Thus, we hypothesize that postbiotics LpD3.5 may elevate mucin levels in the gut which in turn may be associated with reduced gut permeability, inflammation, and better QOL in individuals with IBD.

The LpD3.5 is a common probiotic and has been isolated from human infant gut. This is one of the most common probiotic strains that are listed as Generally Recognized As Safe (GRAS) by the Food and Drug Administration (FDA) and many international lists.

Since L. paracasei is a common probiotic and widely used as a dietary supplement for human consumption. Here, we will use its heat-inactivated form, which is even safer, to determine if its oral consumption changes fundamental biological outcomes such as mucin levels in the gut. These changes may be associated with other physiological but non-clinical outcomes such as gut permeability, inflammation, and QOL in individuals with IBD. This study is planned to address major gaps in knowledge, including the effects of human-origin heat-inactivated postbiotic L. paracasei on the fundamental biology in the gut of individuals with IBD, which may impact their QOL. However, this study is not intended for any commercial purposes, changing labeling, or making medical claims related to L. paracasei. Rather, it is fully academic, aiming to determine the mechanistic action of L. paracasei and decipher ways to modulate gut mucin, permeability, and inflammation, which can aid us in designing future strategies to improve the QOL in individuals with IBD.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older.
2. Individuals with a confirmed diagnosis of IBD, including:

   * History of IBD for more than 3 months
   * Last colonoscopy within 2 years of study entry
   * Mild to moderate IBD symptoms
3. Participants who can provide informed consent with a signature.
4. Body mass index (BMI) between 18 and 40 kg/m²
5. English Speaking

Exclusion Criteria:

Participants meeting any of the following criteria will be excluded:

1. History of severe GI surgery.
2. History of antibiotics, diarrhea, or vomiting within the past 30 days.
3. Use of intravenous corticosteroids within 2 weeks before screening, during screen-ing, or during the study period.
4. Diagnosis with cancer and/or going through chemotherapy/radiation therapy within the past 2 years.
5. Dramatic weight change (>20 pounds) in the past 2 weeks.
6. Using other microbiome-influencing drugs or interventions.
7. Participating in another clinical trial.

11. Ongoing use of non-study probiotics, prebiotics, synbiotics and postbiotics. They can be readmitted if stop such regimens for minimum 30 days.

11.1 Probiotic use is defined as consumption of ≥108 CFU/day, in the form of tablets, capsules, lozenges, powders, or dairy products in which probiot-ics are a major ingredient 12. Heavily consuming (>2 servings per day) yogurt, kefir, kombucha and other fermented food products that can influence microbiome.

13. If they have heart disease, renal disease, active infection, gum bleeding disorder, severe diabetes, obesity (>40 BMI), immunodeficiency, or thyroid disorders.

14. History of anaphylaxis or allergies to probiotics or postbiotics. 15. Uncooperative behavior or any condition that could make the participant potentially non-compliant with the study procedures.

16. Any individuals classified in one of the vulnerable populations, including pregnant women, neonates, prisoners, and children

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-06-15 (Estimated); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Levels of post-intervention fecal mucin (marker of gut barriers) between LpD3.5 and placebo groups | At baseline (pre), 60 days post intervention and 180 days post intervention
  The study determines whether LpD3.5 has any impact on the biological mechanism of mucin that regulates gut permeability. We will analyze whether the dietary grade (heat-killed) LpD3.5 capsule may change the levels of mucin in individuals with inflammatory bowel diseases (IBD).

CONTACTS AND LOCATIONS:
Locations (1):
- University of South Florida, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided